CLINICAL TRIAL: NCT05875792
Title: EvolvRehab - MoveWell Virtual Platform for Stroke Survivors Rapid Rehabilitation Through Fun Exergaming-based Learning
Brief Title: EvolvRehab for Telerehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRIH18P2018
Record Dates: First submitted 2023-02-22; First posted 2023-05-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: telerehabilitation; rehabilitation; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single arm, before and after feasability study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): people who have recently had a stroke and need upper limb rehabilitation
  Interventions: Device: EvolvRehab - MoveWell

INTERVENTIONS:
Device: EvolvRehab - MoveWell — The Intervention has been developed and has a CE mark and has medical device level 1 approvals in the UK. It will be developed with patients in Phase 1 and will consist of initial staff training [training package]. Exercise prescription will be encouraged, in line with usual care, for the either one week (stage 1, phase 2) or six weeks (stage 2, phase 2). Individuals will be able to continue using the EvolvRehab - MoveWell system beyond 6 weeks from stage 2, phase 2, and technical support will continue until the end of the study completion, participants will not be limited in the additional activity that can be performed during this time, and encouraged to do as much as they wish, except if needed for clinical reasons. The intervention will be supported by the clinical team in keeping with routine care. The research therapist will attend clinical visits and support as required. The number of visits will be recorded, and will hopefully reduce to zero over the study.

SUMMARY:
This study includes two stages to develop the use of EvolvRehab telerehabilitation in the use of Stroke patients, early after stroke. All tasks will be conducted by multiple research sites. Stage 2 will include at least 6 weeks of study intervention, and up to 6 months follow-up, where possible.

DETAILED DESCRIPTION:
All tasks in this phase will be conducted by at least two research sites (University of Exeter (site 1) and University of Bristol (site 2)) and the results from stage 1 of the study will be used to inform stage 2, following an amendment to incorporate any changes required.

Stage 1, phase 1: Review of product and processes for the preliminary pilot. The investigators will adopt a Person-Based Approach (user-Centred Design plus behavioural science) to further co-develop/refine the technology and clinical processes for use in National Health Service (NHS) stroke community services (n=15).

Stage 1, phase 2: Iterative pilot. EvolvRehab/MoveWell will be iteratively piloted in five stroke survivors' homes in one NHS team. The investigators will purposefully recruit a heterogeneous sample (e.g. gender, digital literacy, and home context). For this intervention stage of the pilot, patients will give consent. Participants will use EvolvRehab/MoveWell for one week. The research therapist will visit participants' homes alongside research staff to provide support and monitor home safety. A log of issues and feedback will be compiled. We will collect system data to finalise system refinements.

Stage 1, phase 3: Staff focus group. Rehab team staff (clinicians, carers, managers; n = 5) from Site 1 will be convened to agree how EvolvRehab will be deployed in community stroke services. The investigators will identify barriers and facilitators to deployment and report how these will be addressed. This will be advertised via poster which will be sent via email to stakeholders already involved in the study.

Stage 1, phase 4: Service user interviews. Semi-structured interviews will be held with stroke survivors used in stage 1, phase 2 (n=5) to explore issues experienced in using the system in their homes. The investigators will explore support structures (e.g., social networks) and barriers/ facilitators to engagement. Potential changes to software, hardware, support, and training will be mapped and reported. Patient/carer instruction materials will be created. The investigators will create a Digital Inclusion Package. Patients will be contacted to organise this via telephone and/or email.

Stage 1, phase 5: Service specification. A final service and product specification including reference to materials above, will be prepared to inform the second stage of the study.

All tasks in this phase will be conducted by multiple research sites. Stage 2 will include at least 6 weeks of study intervention, and up to 6 months follow-up, where possible.

Stage 2, phase 1: Site engagement and set-up.

At least two sites have expressed firm interest in participating in this study. Site set-up will start at the earliest opportunity, including staff training. Recruitment sites will be rolling, adding additional sites (with appropriate approvals) until the recruitment target is reached.

Stage 2, phase 2: Recruitment and follow-up n = 70. Participants will be identified by their treatment team. Potential participants will be screened against inclusion/ exclusion criteria and read a participant information sheet before consent will be taken. Participants will be shown how to use the system by their treating therapist and provided with additional support as required by the research therapist which will be recorded.

Stage 2, phase 3: Continuation phase n = 70. For the duration of the study, participants will continue to use EvolvRehab as they wish. Use and progression will be recorded by the system. Patients will continue to be provided with support. Support requirements will be logged.

Stage 2, phase 4: Data collection and management n = 70. Outcome Measures will be recorded by a member of the research team, as follows:

Health economic outcomes: Full data for 50 participants

Feasibility of intervention use in stroke services: Full data for 50 participants (Stroke severity and disability); Impairment (motor assessment); physical function (shoulder abduction finger extension, grip strength, barthel); physical activity; communication impairment; Cognitive impairment; Patient activation; Acceptability (amount of use, process interviews, user satisfaction); Safety (adverse events)

Feasibility of potential future clinical trial (Recruitment and retention rate; data completeness)

Clinical effectiveness (Note that this is a single arm study and will not provide definitive evidence of clinical effectiveness). In addition to clinical effectiveness measures. Feasibility of intervention: time in EvolvRehab activities; number of repetitions; health-related quality of life (EQ-5D-5L); carer strain index. Measures of compensation/quality of movement. Subjective reports of effectiveness.

Service utilisation: Measures of utilisation of resources during the study for the health economic analysis (number and duration of staff visits; requirement for technical support; training required).

Stage 2, phase 5: Process interviews n = 15. Interviews with clinicians, participants, and carers post-trial will explore potential improvements and user experience, including testimonials for dissemination. This will be advertised via poster which will be sent via email to stakeholders already involved in the study.

Stage 2, phase 6: Data analysis

Analyses will be conducted under headings:

Health economics (including service utilisation)

Feasibility of delivery (Recruitment and retention rate; data completeness)

Feasibility of future clinical trial: variability of clinical outcomes will allow estimation of sample size for a future trial of system clinical effectiveness. Recruitment and retention rates will be used to estimate necessary recruitment

Clinical effectiveness: analysis will focus on improvement over the course of the study, particularly compensatory movements and disability

Stage 2, phase 7: Dissemination

Dissemination activities will be carried out according to the Dissemination Plan co-written with stroke survivors. The investigators will use a variety of means to disseminate the results to a range of stakeholders. Methods include academic publications and presentations; written reports; articles in publications of stakeholder organisations; presentations to and publications for potential customers. Stakeholders include stroke survivors and the public; health professionals (individuals and organisations); clinical academics; voluntary sector organisations; health and care commissioners and providers.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing motor difficulties in using the paretic arm, with some use of hand/arm as determined by clinical treatment team
* Able to safely participate and complete EvolvRehab activities as determined by clinical treatment team
* Male/female ≥18 years old
* Recently had a stroke requiring upper limb intensive rehabilitation
* The participant is expected to be able to use equipment for a minimum of 1 week
* Capacity to consent to participate
* Able to communicate adequately in English with the research team

Exclusion Criteria:

* Participating in another intervention which the research team deem could interfere with study outcomes
* Any medical condition compromising the safety or the ability to take part to the study as determined by the clinical treatment team (such as insufficient vision or hearing, upper limb condition not linked to stroke, uncontrolled blood pressure, uncontrolled diabetes, co-morbidity)
* History of more than one epileptic seizures since stroke onset or uncontrolled epileptic seizure
* Cognitive or communication impairment such that the participant is unable to follow a two stage command
* Moderate to severe hemi-spatial neglect compromising the ability to take part to the study, as determined by research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment | 6 weeks
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The scale is comprised of five domains and there are 155 items in total:
  Movements are scored between 0 (none), 1 (partial) or 2 (full/ can be elicited) for reflex activity, volitional movement within synergies, volitional movement mixing synergies, volitional movement with little or no synergy, for upper body including wrist and hand.
  Normal reflex activity is scored 0 (hyper), 1 (lively) or 2 (normal).
  Co-ordination is scored 0 (marked), 1 (slight) or 2 (none).
  Sensation is scored 0 (anesthesia), 1 (hypoesthesia or dysesthesia), 2 (normal)
  Joint motion is scored 0 (only few degrees), 1 (decreased), 2 (normal)
  Joint pain is scored 0 (pronounced pain), 1 (some pain), 2 (no pain)

SECONDARY OUTCOMES:
Carer Strain Index (CSI) | 6 weeks
  The CSI can be used to quickly identify families with potential caregiving concerns. It is a 13-question tool that measures strain related to care provision. There is at least one item for each of the following major domains: Employment, Financial, Physical, Social and Time. Positive responses to 7 or more items on the index indicate a greater level of strain. This instrument can be used to assess individuals of any age who have assumed the role of carer for an older adult
Grip strength | 6 weeks
  Hand-grip strength was assessed through the use of a handheld dynamometer. Participants sat with the elbow of the arm which was holding the dynamometer, against the side of their body, and bent to a 90˚ angle. Hand-grip strength was measured three times on each side, with the highest value taken as their maximum grip strength.
European Quality of Life questionnaire (Eq-5D-5L) | 6 weeks
  The measure covers five dimensions of health related quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, scored by level of severity for each dimension (1= no problems, 2= slight problems,3=moderate problems, 4=severe problems, and 5=extreme problems). Overall health status is also measured using a visual analogue score out of 100 whereby higher scores = better quality of life.
The World Health Organization Disability Assessment Schedule (WHODAS) | 6 weeks
  The World Health Organization Disability Assessment Schedule is a generic assessment instrument developed by WHO to provide a standardised method for measuring health and disability across cultures.
Health resource use questionnaire | 6 weeks
  Self-reported questionnaires of healthcare resource utilisation.
Acceptability | 6 weeks
  Questions around: Acceptability of Intervention Measure, Intervention Appropriateness Measure, Feasibility of Intervention Measure.
  Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree
Incidence of adverse events | 6 weeks
  monitoring of any adverse events
System Usability Scale | 6 weeks
  The SUS is a 10 item questionnaire about how easy the rehabkit is to use, with 5 response options (ranging from strongly disagree = 1 to strongly agree 5).
Free-living activity | 6 weeks
  Participants will use bilateral physical activity monitors (accelerometers), which they will wear for up to 8 days prior to the start of the 6-week intervention, to measure a period of "free-living" at baseline and follow-up. This will objectively measure participants' habitual physical activity level. Participants will be asked to continuously wear the monitors for 24 hours a day for up to 8 days.
  The devices will be initialised using the manufactures software under default settings. Alongside this, participants will also be asked to fill out a self-report diary (wake and sleep log) for the days they wear the devices, and if completely necessary, record any time when the devices are removed.
Process interviews | 6 weeks
  Interviews will be led by researchers from UoE. (Interviews with clinicians, participants and carers post-trial will explore potential improvements and user experience, including testimonials for dissemination
Shoulder Abduction Finger extension | 6 weeks
  The SAFE score is calculated by scoring Shoulder Abduction and Finger Extension of the paretic upper limb using the Medical Research Council grades.
  The patient's strength in each of these movements is scored between 0 and 5. 0 = no palpable muscle activity
  1. = palpable muscle activity, but no movement
  2. = limited active range of motion without gravity
  3. = full active range of motion against gravity, but no resistance
  4. = full active range of motion against gravity and resistance, but weaker than the other side
  5. = normal power
Movement quality in "movewell" activities on the EvolvRehab system | 6 weeks
  Number of compensatory movements identified automatically by the EvolvRehab system during prescribed rehabilitation exercises
Movement quantity in "movewell" activities on the EvolvRehab system | 6 weeks
  Measure of how many repetitions of exercises identified automatically by the EvolvRehab system during prescribed rehabilitation exercises
Range of motion | 6 weeks
  Measure of ranges of motion in shoulder flexion, should abduction, elbow flexion (completed on the EvolvRehab system)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Devon and Exeter Hospitals, Exeter, United Kingdom

REFERENCES:
- [Derived] Perks J, McBride P, Mansoubi M, Clatworthy P, Hulme C, Taylor G, Warner M, Dawes H. EvolvRehab-MoveWell telerehabilitation for stroke survivors: study protocol for a feasibility with embedded initial proof-of-concept study. BMJ Open. 2024 May 6;14(5):e078104. doi: 10.1136/bmjopen-2023-078104. PMID 38719328